CLINICAL TRIAL: NCT07312578
Title: A Prospective, Open Label, Randomized Controlled, Phase II Clinical Study of the Combination of Nimotuzumab,Camrelizumab, and Neoadjuvant Chemotherapy in the Treatment of Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Nimotuzumab,Camrelizumab, and Neoadjuvant Chemotherapy（nCT） in the Treatment of Esophageal Squamous Cell Carcinoma
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Department of Digestive Oncology, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nim-ESCC-26
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Nimotuzumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nimotuzumab; camrelizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimotuzumab+Camrelizumab+Neoadjuvant chemotherapy（nCT） (Experimental): Experimental group:
  1. Nimotuzumab: 400mg, Intravenous（iv）, day1（D1）, quaque week（QW）, 6 cycles;
  2. Camrelizumab: 200mg, iv, D1, Q3W, 2 cycles;
  3. Albumin paclitaxel: 125mg/m2, iv, D1, D8, Q3W, 2 cycles;
  4. Cisplatin: 75mg/m2, iv, D1, Q3W, 2 cycles.
  Interventions: Drug: Nimotuzumab; Drug: camrelizumab; Drug: Albumin paclitaxel; Drug: Cisplatin
- Camrelizumab+Neoadjuvant chemotherapy（nCT） (Active Comparator): 1. Camrelizumab: 200mg, iv, D1, Q3W, 2 cycles;
  2. Albumin paclitaxel: 125mg/m2, iv, D1, D8, Q3W, 2 cycles;
  3. Cisplatin: 75mg/m2, iv, D1, Q3W, 2 cycles.
  Interventions: Drug: camrelizumab; Drug: Albumin paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 400mg
  Arms: Nimotuzumab+Camrelizumab+Neoadjuvant chemotherapy（nCT）
Drug: camrelizumab — camrelizumab 200mg
Drug: Albumin paclitaxel — Albumin paclitaxel 125mg/m2
Drug: Cisplatin — Cisplatin 75mg/m2

SUMMARY:
We plan to conduct a single-center,prospective, Open Label, Randomized Controlled, Phase II Clinical Study of the Combination of Nimotuzumab,Camrelizumab, and Neoadjuvant Chemotherapy in the Treatment of Locally Advanced Resectable Esophageal Squamous Cell Carcinoma

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled, open label clinical trial aimed at evaluating the efficacy and safety of the combination of nimotuzumab,camrelizumab, and neoadjuvant chemotherapy in patients with locally advanced resectable esophageal squamous cell carcinoma. The enrolled patients will receive neoadjuvant therapy (camrelizumab ±nimotuzumab+Albumin Paclitaxel+Cisplatin) and esophageal cancer radical surgery (performed within 4 weeks after the last drug treatment). This study includes screening period, treatment period, efficacy follow-up period, and survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

- 1. Sign the informed consent form; 2. Age range: 18-70 years old, both male and female are acceptable; 3. Esophageal squamous cell carcinoma patients diagnosed by histology or cytology; 4.ECOG：0～1； 5. Expected survival period ≥ 12 weeks; 6. Have not received any treatment for primary esophageal tumors in the past, including drug therapy, surgical treatment, and radiation therapy, etc; 7. Clinical staging: cT1-4a, N1-3, M0 (AJCC/UICC esophageal cancer staging (8th edition)), can be surgically resected; 8. Important organ functions meet the following requirements:

1. Absolute neutrophil count ≥ 1.5 × 109, platelet count ≥ 80 × 109, hemoglobin count ≥ 90g/L;
2. Total bilirubin level ≤ 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN (for patients with liver metastases, AST and ALT levels ≤ 5 times ULN);
3. Serum creatinine ≤ 1.5 times ULN or creatinine clearance rate ≥ 60 ml/min (Cockcroft Gault formula);
4. Serum albumin ≥ 28g/L;
5. Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%);
6. Pulmonary function: FEV1/FVC ≥ 70%, FEV1 ≥ 50% normal value, percentage of measured and predicted DLCO (lung diffusion function)>80%.

9. Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, birth control pills, or condoms) during the study period and within 6 months after the end of the study; Within 7 days prior to enrollment in the study, the serum or urine pregnancy test must be negative and the patient must be non lactating; Men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* 1. Patients with any active autoimmune diseases or autoimmune diseases (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; asthma that has been completely relieved in childhood and does not require any intervention in adulthood can be included; asthma that requires medical intervention with bronchodilators cannot be included); 2. The patient is currently using immunosuppressants or systemic hormone therapy to achieve immunosuppression (dose>10mg/day of prednisone or other therapeutic hormones), and has continued to use them within the 2 weeks prior to enrollment; 3. Previously received treatment with EGFR monoclonal antibodies or EGFR tyrosine kinase inhibitors; 4. Patients with any severe and/or uncontrolled illnesses, including:

  1. Patients with poor blood pressure control (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100 mmHg); Suffering from grade I or above myocardial ischemia or infarction, arrhythmia (including QT interval ≥ 480ms), and grade I cardiac dysfunction;
  2. Active or uncontrolled severe infections;
  3. Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA ≥ 104 copies/ml or 2000IU/ml) or hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the detection limit of the analytical method); 5. Patients whose imaging shows that the tumor has invaded important blood vessels or whose researchers have determined that the tumor is highly likely to invade important blood vessels and cause fatal bleeding during subsequent studies; 6. Pregnant or lactating women; Patients with other malignant tumors within 7.5 years (excluding cured skin basal cell carcinoma and cervical carcinoma in situ); 8. Patients with a history of abuse of psychotropic drugs who cannot be quit or those with mental disorders; 9. Patients who have participated in clinical trials of other drugs within the past four weeks; 10. Patients with accompanying diseases that pose a serious threat to patient safety or affect the completion of the study, as determined by the researchers; 11.Researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | up to 2 years
  Pathological complete response (pCR) rate

SECONDARY OUTCOMES:
Event-free survival （EFS） | from enrollment until firstly confirmed and recorded disease progression or death，assessed up to 3 years
  Event-free survival (assessed by the investigator per RECIST v1.1 criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Zhihao MM Lu, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Department of GI Oncology, Peking University Cancer Hospital,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No